CLINICAL TRIAL: NCT03418636
Title: The Staying Safe Intervention: Preventing HCV Among Young Opioid Injectors
Brief Title: The Staying Safe Intervention
Acronym: Ssafe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 652
Record Dates: First submitted 2018-01-12; First posted 2018-02-01 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis C; Opioid Use
Keywords: People who inject drugs; Hepatitis C prevention; Young adults; Behavioral interventions
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staying Safe (Ssafe) (Experimental): Ssafe is delivered in a small group format (consisting of approximately 10-12 participants) by a trained facilitator over 4 2.5-hour sessions (10 hours total). To help promote the maintenance of risk reduction over the trial's 12-month follow-up period, Ssafe participants will be provided with a novel interactive, smartphone-delivered "booster" application based on core Ssafe principles and risk reduction strategies.
  Interventions: Behavioral: Staying Safe (Ssafe)
- Healthy Living (Active Comparator): Healthy Living is a time- and attention-matched control intervention of equivalent session structure and duration as Ssafe (4 2.5-hour sessions; 10 hours total), also delivered in a small group format (10-12 participants). Healthy Living participants will be provided with a publicly available, sleep hygiene-focused smartphone app to promote healthy sleep habits over the trial's follow-up period.
  Interventions: Behavioral: Healthy Living

INTERVENTIONS:
Behavioral: Staying Safe (Ssafe) — Staying Safe motivates and teaches young people who inject drugs (PWID) planning skills and drug use management strategies to enable long-term risk avoidance and the implementation of healthy protective behaviors. Content is presented through guided discussions and role playing exercises, and relies heavily on interactive participation by group members to foster peer-based learning and social reinforcement processes.
  Arms: Staying Safe (Ssafe)
Behavioral: Healthy Living — The content of the Healthy Living intervention is based on the DHHS' Eat Healthy, Be Active Community Workshop curriculum, supplemented with basic sleep hygiene education. Science-based dietary and light physical activity guidelines are demonstrated and promoted to help participants develop and maintain a healthy lifestyle.
  Arms: Healthy Living

SUMMARY:
The growing population of young people who inject drugs (PWID) is at extremely high risk for HCV infection through the use of contaminated injection equipment, yet, to date, no behavioral intervention has been sufficiently potent to produce significant reductions in HCV incidence among PWID. To address this critical public health need, our team developed Staying Safe (Ssafe), an innovative, strengths-based, socio-behavioral HCV prevention intervention found in preliminary research to be highly acceptable and feasible, with strong indications of efficacy. The proposed randomized, controlled trial will assess the effectiveness of the Ssafe intervention in reducing both injection-related HCV/HIV risk behavior and HCV incidence among young adults (ages 18-29) who inject opioids (heroin and/or prescription opioids).

DETAILED DESCRIPTION:
HCV infection is the most common chronic blood-borne infection in the U.S., with the overwhelming majority of new HCV infections occurring among people who inject drugs (PWID). Sharing syringes and other injection equipment is the primary risk factor for HCV transmission. HCV prevalence is extremely high in most U.S. PWID populations (typically ranging from ~40-70%). Research shows that young PWID (under age 30) engage in particularly high rates of risky injection, and that HCV incidence is highest in the first 3-5 years of an individual's injection career. The national significance of this public health problem is heightened by the recent epidemic of prescription opioid (PO) misuse in youth which has evolved into widespread heroin use and injection drug use, creating a new generation of young injectors at risk for HCV (and HIV). These trends demonstrate the urgent need for innovative new approaches to HCV prevention tailored to the growing population of young PWID.

To date, no behavioral intervention has been sufficiently potent to produce significant reductions in HCV incidence in at-risk groups of PWID. To address this critical gap, our team developed Staying Safe (Ssafe), an innovative, strengths-based, socio-behavioral HCV prevention intervention for young PWID. Ssafe addresses multi-level "upstream" determinants of risk that occur relatively early in the causal chain of risk, including eco-social conditions, social relations and risk situations, in addition to directly targeting risky injection practices. Ssafe trains and motivates PWID to better manage drug use in order to avoid situations and practices that promote risky injection (e.g., "binging" on drugs), and to implement health-protective behaviors (e.g., promoting risk-reduction norms in injection networks). In preliminary research we found Ssafe to be highly acceptable and feasible, with strong indications of efficacy.

In this study we propose to conduct a randomized controlled trial to assess the effectiveness of the Ssafe intervention (with a mobile phone-delivered booster application) in reducing injection-related risk behavior and HCV incidence among 18-29 year-olds (n=456) who inject opioids (heroin and/or POs) and test HCV and HIV antibody-negative at baseline. We hypothesize that Ssafe will significantly reduce injection risk behaviors and HCV infections relative to a time- and attention-matched control intervention. We will also examine whether Ssafe's effects are mediated by (a) drug use management practices (injection frequency, overdose, opioid intake, withdrawal episodes); (b) individual-level mechanisms of behavior change (motivation/self-efficacy, planning skills); and (c) key upstream socio-structural and network-level determinants of risk (social support, skills to avoid PWID-associated stigma, drug treatment and SEP utilization, injection network size and risk norms). The proposed trial promises to significantly advance our ability to prevent HCV infection in the growing population of young, PO-initiated injectors.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C antibody-negative
* HIV antibody-negative
* Have injected drugs 4 or more times in the past 30 days
* Current opioid use (verified by rapid urine screen)
* Speak English
* Willing to participate in assigned intervention

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 456 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Injection risk behavior: Syringe-sharing | 3 months
  number of times receptively shared syringes
Injection risk behavior: Syringe-sharing partners | 3 months
  number of people receptively shared syringes with
Injection risk behavior: Secondary injection equipment-sharing | 3 months
  number of times receptively shared secondary injection equipment (including cookers, cottons, water and water containers combined)
Injection risk behavior: Secondary injection equipment-sharing partners | 3 months
  number of people receptively shared secondary injection equipment with (including cookers, cottons, water and water containers combined)
Injection risk behavior: Backloading | 3 months
  number of times backloaded
Injection risk behavior: Backloading partners | 3 months
  number of people backloaded with

SECONDARY OUTCOMES:
Hepatitis C incidence | 12 months
  hepatitis C antibody-positive rapid test result (OraQuick)
Overdose events | 3 months
  opioid-related episodes involving loss of consciousness, non-responsiveness and/or administration of naloxone
Injection frequency | 30 days
  average number of daily and monthly injections
Injection-related complications | 3 months
  number and type of physical complications from injection drug use

OTHER OUTCOMES:
Injection network size | 3 months
  number of people injected with (i.e., in the presence of these people)
Motivation/Self-efficacy to inject safely and manage opioid intake | 3 months
  Total score on the Staying Safe Self-Efficacy Scale (8 items; possible score range = 0-32), an investigator-developed and validated instrument (Mateu-Gelabert et al., 2014).
OUD treatment participation | 3 months
  participation in Medication-Assisted Treatment (MAT) for Opioid Use Disorder (OUD)
Opioid withdrawal | 3 months
  frequency of opioid withdrawal episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Staying Safe Study 235 Eldridge Street, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided